CLINICAL TRIAL: NCT05937672
Title: Cold Atmospheric Plasma Device for the Treatment of Molluscum Contagiosum and Verruca Vulgaris in Pediatric Patients - Open-Label Extension Study
Brief Title: Cold Atmospheric Plasma Device Extension Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: The Skin Center Dermatology Group (Industry)
Responsible Party: Principal Investigator, Lara Wine Lee, Assistant Professor, Dermatology and Dermatologic Surgery, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00127338
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-01

CONDITIONS: Verruca Vulgaris; Molluscum Contagiosum
Keywords: Plasma; Warts; Molluscum; Pediatric; Dermatology
MeSH Terms: conditions — Warts; Molluscum Contagiosum

STUDY DESIGN:
Intervention Model Description: This is an open-label extension study. During a clinical care visit, if a patient is eligible and agrees to participate, lesions will be selected by the dermatologist prior to procedure. All lesions selected will be treated with non-thermal atmospheric plasma (NTAP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cold Atmospheric Plasma (CAP) (Experimental): We are proposing an open-label extension study of a floating electrode-dielectric barrier device (FE-DBD), a Cold Atmospheric Plasma (CAP) device for the treatment of Verrucae Vulgaris and Molluscum Contagiosum. While novel to the medical field, and especially to dermatology, there are already a number of publications regarding its use on human skin in adults and children. CAP devices utilize noble gases (such as helium) to deliver plasma state matter to the skin. As its name implies, the generated plasma stream is of near skin temperature and it exists on normal atmospheric pressure. During the generation of the plasma there is no electric contact with the patient. The treatment does not increase skin surface temperature and the used helium gas, the same as used for balloons, being a noble gas does not cause a chemical reaction with the skin. The flow of the gas is slow, thus there is no mechanical effect on the skin.
  Interventions: Device: Floating electrode-dielectric barrier device (FE-DBD) cold atmospheric plasma (CAP)

INTERVENTIONS:
Device: Floating electrode-dielectric barrier device (FE-DBD) cold atmospheric plasma (CAP) — The treatment device in this study generates cold atmospheric plasma. Cold atmospheric plasma has certain properties of plasma, such as ionized gas molecules. To create plasma, a pulse generator supplying 20 kilovolt pulse of 20-ns pulse width at 200 Hz (FPG10-01NM10, FID GmbH, Burbach, Germany) to a 5-mm diameter quartz-covered copper electrode of 10-cm length and 1 - 13mm quartz thickness. These nanosecond pulse parameters were chosen to provide sufficient treatment dose at the high level of plasma uniformity required to avoid any tissue damage. We will treat the lesions for approximately 1 to 2 minutes each, moving the electrode gently over the treatment area.
  Other Names: Non-thermal atmospheric pressure plasma (NTAP)

SUMMARY:
Patients between 4-21 years of age with at least one wart or molluscum lesion are eligible to participate in this study. The duration of the study is a minimum of 4 weeks with the maximum duration of monthly treatments for one year, depending on lesion clearance. The number of lesions will be chosen by the dermatologist. Patients who opt to participate will receive non-thermal, or cold, atmospheric plasma to treat all lesions selected. Safety profile as well as changes in size, pain and appearance will be measured. Photographs and dermatologist impressions will be used to measure treatment response.

ELIGIBILITY:
Inclusion Criteria:

* All patients from 4-21 years old with at least 1 lesion of vercurra or molluscum.
* Willingness of the participant and their guardian to provide consent when applicable.

Exclusion Criteria:

* Unwillingness to participate in the study
* Received any treatment on the lesion in the past month determined by review of their medical record
* Immunodeficiency determined by review of their medical record.
* Adverse response to prior treatments determined by review of medical record.
* Signs of self-resolution determined by study team members.
* Conditions that lead to excessive scarring determined by study team members.
* Face and genital lesions determined by study team members.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of lesions with no response | Maximum of 12 months
  Absence of change in appearance of targeted lesion. Molluscum is defined as the visualization of a central umbilication with polylobular, white to yellow, amorphous structures. A peripheral crown of radiating or punctiform vessels may also be present. Warts are defined as grouped papillae, with dotted or loop vessels, and/or hemorrhagic points and lines often surrounded by a whitish halo.
Number of lesions with partial response | Maximum of 12 months
  There is change in the size, dyspigmentation, or discomfort of the targeted lesion as compared to its appearance and symptoms at the initial visit, but the lesion remains grossly visible. Molluscum is defined as the visualization of a central umbilication with polylobular, white to yellow, amorphous structures. A peripheral crown of radiating or punctiform vessels may also be present. Warts are defined as grouped papillae, with dotted or loop vessels, and/or hemorrhagic points and lines often surrounded by a whitish halo. Changes in the characteristics of the targeted lesions will be evaluated by a dermatologist and documented via photographs at follow-up visits at 4, 8, and 12 weeks, with the final outcome measured at the 12-week visit.
Number of lesions with complete response | Maximum of 12 months
  Targeted lesion is no longer grossly visible.
Number of treatments to complete lesion resolution | Maximum of 12 months
  Comparing number of treatments necessary for complete response.

SECONDARY OUTCOMES:
Adverse events from CAP tolerability questionnaire | Maximum of 12 months
  This questionnaire measures tolerability of cold atmospheric plasma treatment. Assessment of dryness, peeling, scaling, erythema, edema, stinging, burning sensation, itching, scarring and dyspigmentation will each be assessed individually by means of a standardized grading scale (0 = absent; 1 = mild; 2 = moderate; 3 = severe)
Average score of visual analogue scale associated with treatment | Maximum of 12 months
  The visual analogue scale (VAS) is a validated subjective measurement of pain experienced by the patient. It consists of visual-numeric scale, numbered from 0-10. (0) indicate absence of pain or "no pain at all", while (10) indicates severe pain or "worst imaginable pain". This is supplemented by six faces with different expressions, ranging from happy to extremely upset. Each facial expression is assigned a numerical scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No